CLINICAL TRIAL: NCT07171853
Title: The Carbon Footprint Study of Colonoscopy for Colorectal Cancer Screening and Various Techniques of Colonic Polypectomy
Brief Title: The Carbon Footprint Study of Colonoscopy
Status: Recruiting | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Assoc. Prof. Dr., King Chulalongkorn Memorial Hospital
Other Study IDs: RP028
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy
Keywords: Carbon footprint; Colonoscopy; Colonic polypectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic Colonoscopy: Patient receiving diagnostic colonoscopy for colorectal cancer screening without therapeutic intervention
- Colonoscopy with colonic polypectomy: Patient receiving colonoscopy with various techniques of colonic polypectomy

SUMMARY:
With global warming intensifying, GI endoscopy is among the top three greenhouse gas-emitting medical procedures. Colonoscopy, a cornerstone for colorectal cancer (CRC) screening, significantly contributes to the carbon footprint (CF). This study quantifies CO₂ emissions in different steps of colonoscopy and evaluates the environmental impact of common polypectomy techniques to establish baseline CF data and identify opportunities for mitigation. This study included patients undergoing colonoscopy for CRC screening. CO₂ emissions were comprehensively measured at each step of the procedure (pre-, during, and post-colonoscopy), including energy consumption, all equipment and medications, waste management, and endoscopy reprocessing. Emission data were also collected for common polypectomy techniques, including cold forceps biopsy (CFB), cold snare polypectomy (CSP), hot snare polypectomy (HSP), and hot snare endoscopic mucosal resection (EMR), all performed according to standard polypectomy protocols.

DETAILED DESCRIPTION:
Global warming refers to the long-term increase in Earth's average surface temperature, primarily caused by the buildup of greenhouse gases in the atmosphere due to human activities. The carbon footprint of a colonoscopy refers to the total greenhouse gas emissions (primarily CO₂ equivalents) generated throughout the procedure. While colonoscopy for colon cancer screening improves survival outcomes, it still contributes to environmental impact through energy use, medical supplies, and waste. Calculating a carbon footprint involves estimating the total greenhouse gas emissions, usually expressed in carbon dioxide equivalents (CO₂e).

Main formula : Carbon footprint (CO₂e) = Activity Data × Emission Factor

Carbon footprint assessment is a tool for assessing the magnitude of greenhouse gas emissions from public health care processes for planning, developing and systematically improving public health systems to reduce carbon footprints leading to environmental sustainability.

Carbon footprint measurement in this study

1. Volunteers underwent bowel preparation by taking laxatives until their stool appearance met the clear criteria. The amount of laxative taken was recorded.
2. A nurse conducted a medical history interview using a standardized safety checklist before the colonoscopy, measured the patient's vital signs, and established intravenous access for administering medication or fluids.
3. Research participants were fitted with a nasal oxygen delivery device and given intravenous sedatives to induce an appropriate level of sedation. Vital signs and fingertip oxygen saturation levels were monitored before starting the colonoscopy.
4. During the colonoscopy, the nurse monitored vital signs and oxygen saturation periodically and adjusted the sedative dosage based on the patient's level of consciousness.
5. Patients underwent colonoscopy for colorectal cancer screening and diagnosis. If a colonic polyp was found, it was removed according to clinical indications and current treatment guidelines. The size of the polyp was estimated visually by comparing it with the size of the resection instrument. In the event of bleeding or perforation, endoscopic procedures were performed as indicated for treatment. During the procedure, all equipment used, the volume of water, the type and amount of sedative medication, and the duration of the colonoscopy and colonic polypectomy were recorded for subsequent carbon footprint analysis.
6. The removed colonic polyp tissue was preserved in a formalin-containing specimen jar for pathological examination by a pathologist.
7. After the colonoscopy, the patient was transferred to a recovery room, where vital signs were monitored periodically until the participant regained full consciousness.
8. After polypectomy, the patient resumed antiplatelet and anticoagulant medications according to the timing recommended by standard clinical guidelines.

The data from the patient's intake of laxatives for bowel preparation through to the completion of the colonoscope cleaning process was recorded and analyzed to calculate the carbon footprint in collaboration with the faculty team from the Environmental Research Institute of Chulalongkorn University.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years

Exclusion Criteria:

* Patient status grade III-V according to the American Society of Anesthesiologists (ASA)
* Poor bowel preparation (grade <6 in the Boston Bowel Preparation Scale [BBPS])
* Endoscopic JNET type III or suspicion of malignancy
* Hematologic or coagulation disorders, Plt<140,000/mcL, INR>1.5
* anti-platelet/anticoagulant medication that could not be paused as recommended in the current guideline
* Emergency colonoscopy, GI bleeding, unstable vital sign, critical ill patient
* Inflammatory bowel disease
* Pregnancy
* Severe cardiopulmonary disease
* Severe infection
* Malignancy
* History of allergy to IV sedative medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years who received a colonoscopy at King Chulalongkorn Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Carbon footprint of colonoscopy for colorectal cancer screening and various techniques of colonic polypectomy | 4 months after start this study
  To calculate carbon footprint from colonoscopy for colorectal cancer screening and various techniques of colonic polypectomy

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Steubing B, de Koning A, Merciai S, Tukker A. How do carbon footprints from LCA and EEIOA databases compare? A comparison of ecoinvent and EXIOBASE. Journal of Industrial Ecology. 2022;26(4):1406-22.
- [Background] Turner DA, Williams ID, Kemp S. Greenhouse gas emission factors for recycling of source-segregated waste materials. Resources, Conservation and Recycling. 2015;105:186-97.
- [Background] McGinnis S, Johnson-Privitera C, Nunziato JD, Wohlford S. Environmental Life Cycle Assessment in Medical Practice: A User's Guide. Obstet Gynecol Surv. 2021 Jul;76(7):417-428. doi: 10.1097/OGX.0000000000000906. PMID 34324694
- [Background] Sevigne-Itoiz E, Mwabonje O, Panoutsou C, Woods J. Life cycle assessment (LCA): informing the development of a sustainable circular bioeconomy? Philos Trans A Math Phys Eng Sci. 2021 Sep 20;379(2206):20200352. doi: 10.1098/rsta.2020.0352. Epub 2021 Aug 2. PMID 34334023
- [Background] Yu X, Tan C. China's process-related greenhouse gas emission dataset 1990-2020. Sci Data. 2023 Jan 25;10(1):55. doi: 10.1038/s41597-023-01957-y. PMID 36697420
- [Background] Rodriguez de Santiago E, Dinis-Ribeiro M, Pohl H, Agrawal D, Arvanitakis M, Baddeley R, Bak E, Bhandari P, Bretthauer M, Burga P, Donnelly L, Eickhoff A, Hayee B, Kaminski MF, Karlovic K, Lorenzo-Zuniga V, Pellise M, Pioche M, Siau K, Siersema PD, Stableforth W, Tham TC, Triantafyllou K, Tringali A, Veitch A, Voiosu AM, Webster GJ, Vienne A, Beilenhoff U, Bisschops R, Hassan C, Gralnek IM, Messmann H. Reducing the environmental footprint of gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) and European Society of Gastroenterology and Endoscopy Nurses and Associates (ESGENA) Position Statement. Endoscopy. 2022 Aug;54(8):797-826. doi: 10.1055/a-1859-3726. Epub 2022 Jul 8. PMID 35803275
- [Background] Vaccari M, Tudor T, Perteghella A. Costs associated with the management of waste from healthcare facilities: An analysis at national and site level. Waste Manag Res. 2018 Jan;36(1):39-47. doi: 10.1177/0734242X17739968. Epub 2017 Nov 14. PMID 29132259
- [Background] Ferlitsch M, Hassan C, Bisschops R, Bhandari P, Dinis-Ribeiro M, Risio M, Paspatis GA, Moss A, Libanio D, Lorenzo-Zuniga V, Voiosu AM, Rutter MD, Pellise M, Moons LMG, Probst A, Awadie H, Amato A, Takeuchi Y, Repici A, Rahmi G, Koecklin HU, Albeniz E, Rockenbauer LM, Waldmann E, Messmann H, Triantafyllou K, Jover R, Gralnek IM, Dekker E, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2024. Endoscopy. 2024 Jul;56(7):516-545. doi: 10.1055/a-2304-3219. Epub 2024 Apr 26. PMID 38670139
- [Background] Iwatate M, Sano Y, Tanaka S, Kudo SE, Saito S, Matsuda T, Wada Y, Fujii T, Ikematsu H, Uraoka T, Kobayashi N, Nakamura H, Hotta K, Horimatsu T, Sakamoto N, Fu KI, Tsuruta O, Kawano H, Kashida H, Takeuchi Y, Machida H, Kusaka T, Yoshida N, Hirata I, Terai T, Yamano HO, Nakajima T, Sakamoto T, Yamaguchi Y, Tamai N, Nakano N, Hayashi N, Oka S, Ishikawa H, Murakami Y, Yoshida S, Saito Y; Japan NBI Expert Team (JNET). Validation study for development of the Japan NBI Expert Team classification of colorectal lesions. Dig Endosc. 2018 Sep;30(5):642-651. doi: 10.1111/den.13065. Epub 2018 Jun 26. PMID 29603399
- [Background] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Background] ASGE Standards of Practice Committee; Early DS, Ben-Menachem T, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Jain R, Jue TL, Khan KM, Malpas PM, Maple JT, Sharaf RS, Dominitz JA, Cash BD. Appropriate use of GI endoscopy. Gastrointest Endosc. 2012 Jun;75(6):1127-31. doi: 10.1016/j.gie.2012.01.011. No abstract available. PMID 22624807
- [Background] Cunha Neves JA, Rodriguez de Santiago E, Aabakken L. Approaches for greening endoscopy and reducing waste. Gut. 2023 Nov 24;72(12):2204-2206. doi: 10.1136/gutjnl-2023-330917. No abstract available. PMID 37977580
- [Background] Brown JJ, Asumeng CK, Greenwald D, Weissman M, Zauber A, Striplin J, Weng O, List JM, Farley SM, Winawer SJ. Decreased colorectal cancer incidence and mortality in a diverse urban population with increased colonoscopy screening. BMC Public Health. 2021 Jun 30;21(1):1280. doi: 10.1186/s12889-021-11330-6. PMID 34193094
- [Background] Doubeni CA, Corley DA, Quinn VP, Jensen CD, Zauber AG, Goodman M, Johnson JR, Mehta SJ, Becerra TA, Zhao WK, Schottinger J, Doria-Rose VP, Levin TR, Weiss NS, Fletcher RH. Effectiveness of screening colonoscopy in reducing the risk of death from right and left colon cancer: a large community-based study. Gut. 2018 Feb;67(2):291-298. doi: 10.1136/gutjnl-2016-312712. Epub 2016 Oct 12. PMID 27733426
- [Background] Han J, Tan Z, Chen M, Zhao L, Yang L, Chen S. Carbon Footprint Research Based on Input-Output Model-A Global Scientometric Visualization Analysis. Int J Environ Res Public Health. 2022 Sep 9;19(18):11343. doi: 10.3390/ijerph191811343. PMID 36141618
- [Background] Maurice JB, Rochford A, Marshall S, Sebastian S, Dhar A, Hayee B; Green Endoscopy group. Green endoscopy: using quality improvement to develop sustainable practice. Frontline Gastroenterol. 2021 Jun 7;13(4):342-345. doi: 10.1136/flgastro-2021-101874. eCollection 2022. No abstract available. PMID 35722605
- [Background] Park SB, Cha JM. Gastrointestinal endoscopy's carbon footprint. Clin Endosc. 2023 May;56(3):263-267. doi: 10.5946/ce.2023.003. Epub 2023 Mar 31. PMID 36997185
- [Background] Lacroute J, Marcantoni J, Petitot S, Weber J, Levy P, Dirrenberger B, Tchoumak I, Baron M, Gibert S, Marguerite S, Huppertz J, Gronier O, Derlon A. The carbon footprint of ambulatory gastrointestinal endoscopy. Endoscopy. 2023 Oct;55(10):918-926. doi: 10.1055/a-2088-4062. Epub 2023 May 8. PMID 37156511
- [Background] Purohit A, Smith J, Hibble A. Does telemedicine reduce the carbon footprint of healthcare? A systematic review. Future Healthc J. 2021 Mar;8(1):e85-e91. doi: 10.7861/fhj.2020-0080. PMID 33791483
- [Background] Zandalinas SI, Fritschi FB, Mittler R. Global Warming, Climate Change, and Environmental Pollution: Recipe for a Multifactorial Stress Combination Disaster. Trends Plant Sci. 2021 Jun;26(6):588-599. doi: 10.1016/j.tplants.2021.02.011. Epub 2021 Mar 18. PMID 33745784
- [Background] https://www.who.int/news-room/fact-sheets/detail/climate-change-and-health.
- [Background] Information NNCfE. Monthly global climate report for annual 2022. NOAA Washington, DC; 2023.